CLINICAL TRIAL: NCT05490966
Title: Effects of Isometric Muscle Fatigue on Trunk Muscle Stiffness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Primorska (Other)
Responsible Party: Principal Investigator, MatejVoglar, Assistant Professor, PhD, University of Primorska
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SWE_Isometric
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Muscle Tightness
Keywords: multifidus; erector spinae; muscle stiffness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Isometric fatigue (Experimental): Fatiguing intermittent isometric exertions of trunk extensor muscles will be performed.
  Interventions: Other: isometric trunk extensor muscles fatigue

INTERVENTIONS:
Other: isometric trunk extensor muscles fatigue — Participants will perform three sets of intermittent isometric efforts between 50 and 60 percents of their maximal isometric strength. A padded force sensor will be placed approximately at the level of the 7th thoracic vertebrae. The first two sets will last six minutes each, while the third set will last three minutes. Between each set participants will rest for two minutes.

SUMMARY:
Interventional study of the effects of a trunk extensor muscles fatigue protocol on trunk extensors stiffness.

DETAILED DESCRIPTION:
Single visit interventional study of the effects of a trunk extensor muscles fatigue protocol on multifidus and erector spinae muscle stiffness measured by Ultrasound based Shearwave elastography.

ELIGIBILITY:
Inclusion Criteria:

* Physically active at least 3 hours a week

Exclusion Criteria:

* Low back pain in the past 6 months
* History of chronic low back pain
* History of spinal or pelvic operation
* Hypermobility, more than 4 points on Beighton scale
* Cardiovascular or systemic diseases
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2022-09-10 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-18 (Actual)

PRIMARY OUTCOMES:
Change of trunk extensors muscle stiffness | 1 hour
  Muscle stiffness will be measured at rest and during standardised sub-maximal exertions in prone lying position. Muscle stiffness will be expressed as the shear modulus value in kilopascals.

SECONDARY OUTCOMES:
Change of muscle electromyography mean amplitude | 1 hour
  Muscle activation of trunk extensors will be measured using superficial electromyography at rest and during two standardised sub-maximal exertions in prone lying position (single arm raise and upper body raise). Mean amplitude in six to eight second time frames will be calculated.

OTHER OUTCOMES:
Change in lumbar range of motion | 1 hour
  Lumbar range of motion will be evaluated using Modified modified Schober test.

CONTACTS AND LOCATIONS:
Overall Officials: Matej Voglar, PhD, Principal Investigator — University of Primorska, Faculty of Health Sciences
Locations (1):
- University of Primorska, Faculty of Health Sciences, Izola, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
Coded individual dat will be uploaded on public scientific data repository
Supporting Information: Study Protocol